CLINICAL TRIAL: NCT04077086
Title: SWISH (See Well to Stay In ScHool): Randomised Trial of Spectacle Distribution to Secondary School Children With Myopia to Increase Academic High School Attendance Rates in Rural Communities)
Brief Title: Correcting Myopia Among Secondary School Children to Increase Academic High School Attendance Rates in Rural Communities
Acronym: SWISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other); Stanford University (Other); New England College of Optometry (Other); Clearly (Other); Ningxia Medical University (Other); He Eye Hospital (Other); He University (Other)
Responsible Party: Principal Investigator, Nathan Congdon, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MR/S023208/1
Record Dates: First submitted 2019-08-07; First posted 2019-09-04 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Refractive Errors
Keywords: Refractive error; Myopia; Academic high school attendance; Education attainment; Spectacle wear compliance; Mental health well-being; Progression of shortsightedness
MeSH Terms: conditions — Refractive Errors; Myopia | interventions — Eyeglasses

STUDY DESIGN:
Intervention Model Description: Children in Year 1 at 111 randomly-selected middle-schools in Liaoning, northern China, will be randomized by school to receive free glasses and a teacher-based incentive to promote wear, or prescriptions only.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study personnel assessing trial outcomes will be masked as to children's study group assignment, which will be simplified by the fact that there will be participants with and without glasses at both Intervention and Control schools. It is not ethical in this setting to provide Control participants with placebo treatment (glasses with zero power lenses), but students, parents and teachers will not be informed of either the overall design of the study or the explicit treatment intervention assignment. Only one school will be selected in each township, minimizing the possibility of cross arm communication and contamination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Children at Intervention schools will receive free spectacles of a design they select, based on the child's measured refractive power and dispensed at school by the study optometrist. Additionally, teachers (but not children) in eligible classes will be informed that if 80% spectacle compliance as measured across three separate unannounced inspections was achieved, they will be given an incentive of an conditional cash transfer. The cash transfer will be deposited into the teacher's bank accounts directly.
  Interventions: Device: Spectacles
- Control (No Intervention): Children at Control schools will receive a glasses prescription and letter to the parents informing them of the refractive status of their child, with free glasses provided only at the end of the trial. No teacher incentive will be offered. Service offered to the Control group exceeds standard care, in that no school-based programs of vision screening and refraction currently exist in the study area, or in most of rural China.

INTERVENTIONS:
Device: Spectacles — Intervention group children in middle school Year 1 will receive spectacles in December 2024. Assuming that the relevant effects of treatment (glasses wear) on the main study outcome are complete once examinations determining high school attendance are finished at the end of Middle School Year 3, Intervention participants will have undergone 32 months (December 2024 - July 2027) of treatment by the endpoint of the trial.
  Other Names: Glasses
  Arms: Intervention

SUMMARY:
Chinese children are some of the most short-sighted in the world, but only one in five children in poor areas who needs glasses has them. Our team has already shown in other trials that giving children free glasses leads to better grades and that free glasses have a bigger impact on grades than factors like parents' education level and the amount of money a family has. The effect on grades from glasses is greater than from other health services in school, like giving vitamins. Only about one in three children in rural China goes on to a regular, non-vocational high school. The investigators would like to show the Chinese government strong evidence of what glasses can do to help children continue their education, in order to help convince the government to carry out national programs to provide free glasses for children who need them.

Study Plan: The investigators will choose 111 middle schools at random in Liaoning, northern China, and all children in Year 1 at each school will go at random into one of two groups: either a group getting free glasses, with support from teachers to push them to wear the glasses ("Intervention") or a group getting just glasses prescriptions ("Control.") The main study outcome will be the proportion of children going on to academic (as opposed to vocational) high school, and the study is powered to detect a 10% difference in this figure between groups.The study will also assess whether children wear their glasses at school and how often they use blackboards (which disadvantage short-sighted children) vs textbooks to learn from. These other outcomes will help us to better understand the causal pathway between vision and high school attendance. We will also study the total cost of providing glasses and the teacher support to wear them per additional student attending academic high school, as well as student mental health outcomes. We will also collect data on the progression of nearsightedness. The hypothesis of this study is that providing glasses will increase academic high school attendance.

DETAILED DESCRIPTION:
Research question: Will providing free glasses to myopic rural Chinese students, with a teacher incentive to promote use, increase academic high school attendance?

Design: Cluster-randomised controlled trial

Rationale: Rural Chinese children have high myopia prevalence, but poor access to glasses. Our previous trials show giving free glasses significantly improves academic performance, with greater effect size than parental education or family income, equaling or exceeding other classroom-based medical interventions. Non-vocational (academic) high school attendance is only 30% in rural western China. Strong evidence of educational benefit from glasses is needed to spur adoption of national distribution programs.

Methods: Children in Year 1 at 111 randomly-selected middle schools in Liaoning, Northern China, will be randomized by school to receive free glasses and a trial-proven teacher-based incentive to promote wear (Intervention) or prescriptions only (Control). The main outcome 3 years later will be high school attendance (powered to detect 10% difference between study groups); secondary outcomes of compliance and use of near versus distance classroom learning aids will elucidate biological plausibility of a causal pathway between myopia correction and learning. Local knowledge and attitudes about myopia and spectacle use and intervention cost-effectiveness will be studied.

Statistical methods to be employed in the analysis and justification for the choice of sample size:

Adjusted- and unadjusted-comparison of the difference between study groups

Principal analyses for the main trial will include:

* Of attendance at academic high school after Year 3 of middle school (as opposed to following a vocational pathway or leaving school).
* of observed spectacle wear at un-announced examinations at school and for self-efficacy scores.
* of mental health outcomes after Year 1 year of intervention

Sample size: Assuming 120 students per school undergoing vision screening, 50% of children failing vision screening, 30% of these needing glasses, α=0.05, intra-class correlation=0.10, explained variation by covariates=0.40, difference between the groups in the main study outcome=10%, high-school attendance rate in the Control group=50%, a sample size of 111 middle-schools (55 or 56 in each group) will provide power=80%.

Loss to follow-up in our previous school-based trials in China, SWLW I and II, was approximately 4% over the course of one school year, and so our calculations here assume a loss to follow-up of 10% over 2-3 years. However, we have not adjusted for non-compliance because we will use a strict intention-to-treat analytic approach where children in schools allocated to the Intervention group will be analysed as such irrespective of compliance and because our intention is to test the policy of making free glasses available to those students who need them, rather than the effect of those students actually wearing the glasses. Further, our expected effect size is based conservatively on previous trials with compliance rates of approximately 40%, which we feel can be improved on in the current trial with teacher incentives as above.

ELIGIBILITY:
Inclusion Criteria:

* Year 1 classes (likely age 12-13 years) at the recruited schools
* Have uncorrected (without glasses) visual acuity of ≤6/12 in both eyes;
* Refractive error meets cut-offs shown to be associated with significantly greater improvement in visual acuity when corrected (myopia ≤-0.75 diopters (D, or astigmatism (non-spherical refractive error) ≥1.00 D);
* Visual acuity can be improved to >= 6/7.5 in at least one eye with glasses.

Exclusion Criteria:

* Presence of visually-significant ocular condition besides refractive error

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10000 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Academic high school attendance | In July following completion of Year 3 of Middle School. This occurs after 32 months of participant followup.
  Proportion of children who continue to academic high school as opposed to vocational high school or no additional schooling, assessed by systematically contacting parents, teachers and students to ascertain enrolment status

SECONDARY OUTCOMES:
Compliance with spectacle wear | After 12 months of participant followup
  Actual presence of spectacles on the child's face (rather than having glasses at school) at the time of an unannounced examination.
Blackboard use | After 12 months of participant followup
  Frequency of blackboard versus textbook use in the major subjects (Maths, Chinese, English) on a questionnaire administered to teachers, and answered as "all", "most", "about half", little" or "none" of teaching.
Cost effectiveness of intervention. | At study closeout, after 32 months of participant followup
  Calculated as ratio of incremental cost to proportion of children who continue to academic high school as opposed to vocational high school or no schooling. Incremental cost is the difference of costs between implementation of intervention and control. Intervention costs will comprise the screening test, glasses (including replacements) and teacher incentives.
Depression and Anxiety | At baseline and 12 months post-treatment
  Depression and anxiety score measured with Anxiety Stress Scale (DASS). The score range for depression, anxiety and stress are 0-42, with higher score indicates more severe mental health problems.
Self Esteem | At baseline and 12 months post-treatment
  Self-esteem score measured with the Rosenberg Self-esteem Scale. The scores range from 0-30, with higher scores indicate higher self-esteem.
Emotional and behavioral problems | At baseline and 12 months post-treatment
  Emotional and behavioral problems score using the Strengths and Difficulties Questionnaire (SDQ), with difficulties score ranges from 0 to 40, Prosocial scale ranges from 0-10, with higher score indicates severe mental health and behavioral problems.
Parent-proxy quality of life | At baseline and 12 months post-treatment
  Parent-proxy quality of life will be measured by using Pediatric Quality of Life Inventory™ Generic Core Scales, with scores range from 0-100. The higher score, the better the quality of life
Progression of Shortsightedness | At baseline and 12 months post-treatment
  Progression of Shortsightedness will be measured using change in refraction over time

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD, MPH, Principal Investigator — Queen's University, Belfast
Locations (3):
- China (2):
  - He Eye Specialist Hospital, Shenyang, Liaoning
  - Ningxia University, Yinchuan, Xixia
- Centre for Public Health, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No